CLINICAL TRIAL: NCT00901394
Title: Influence of Preoperative Vitamin B12 and Folate Administration on Homocysteine Concentrations After Nitrous Oxide Anesthesia
Brief Title: Vitamin B12 and Folate Administration on Homocysteine Concentrations After Nitrous Oxide Anesthesia
Acronym: Mini-VINO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Foundation for Anesthesia Education and Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 09-0074
Record Dates: First submitted 2009-05-08; First posted 2009-05-13 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Cardiovascular Abnormalities
Keywords: Nitrous oxide; cobalamin; homocysteine; vitamin B12; folate; No specific diseases targeted
MeSH Terms: conditions — Cardiovascular Abnormalities | interventions — Nitrous Oxide; Sodium Chloride; nitrox; Air

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment 1 (Experimental): B12-Folic acid, nitrous oxide
  Interventions: Drug: B12-Folic Acid, nitrous oxide; Drug: Nitrous oxide (NO) and placebo
- Treatment 2 (Active Comparator): Nitrous oxide (NO) and placebo
  Interventions: Drug: Nitrous oxide (NO) and placebo; Other: Placebo
- Control group (Placebo Comparator): oxygen nitrogen
  Interventions: Other: Placebo; Other: oxygen nitrogen

INTERVENTIONS:
Drug: B12-Folic Acid, nitrous oxide — IV vitamin B12 (cyanocobalamin) 1 mg, single administration over 30 min.
  IV folic acid, 5 mg, single administration over 30 min.
  Both diluted in 250 ml normal saline.
  Other Names: b supplements
  Arms: Treatment 1
Drug: Nitrous oxide (NO) and placebo — 60% nitrous oxide anesthesia plus saline
  Other Names: nitrous oxide
  Arms: Treatment 1; Treatment 2
Other: Placebo — Saline
  Other Names: saline
  Arms: Control group; Treatment 2
Other: oxygen nitrogen — 60% air and oxygen mix.
  Other Names: air
  Arms: Control group

SUMMARY:
The goal of this study is to find out if giving intravenous B-vitamins before general anesthesia with nitrous oxide prevents the increase in homocysteine, a metabolite that has been linked to cardiovascular complications.

DETAILED DESCRIPTION:
Patients will be randomized into the following arms:

* Arm A: patients will receive N2O (60% N2O/40% O2) in an open-label fashion during surgery and vitamin supplementation (vitamin B12, 1 mg, and folate, 5 mg) before surgery.
* Arm B: patients will receive N2O 60% N2O/40% O2) in an open-label fashion during surgery and placebo before and after surgery.
* Arm C: patients will not receive N2O, vitamin supplementation, or placebo during/before surgery. Patients in this arm will not be randomized.

Patients will have blood drawn (total of 1-2 teaspoons over 3 days). We will take these samples before their surgery, when their surgery is completed, and in the morning of post-operative day 1. We will be checking their troponin I and troponin T, homocysteine, Vitamin B12, and folate levels. We will also perform a 12-lead EKG. Before and after surgery for patients in Arm A or B, will receive either vitamin B12 (1 mg) and folic acid (5 mg) (or placebo) added to their IV infusion. We also plan to use a non-invasive test known as a nerve conduction study to measure the function of their nerve system. Briefly, 2 small electrodes are attached to their skin over a nerve and, like an EKG, faint electrical pulses are generated and recorded. A typical nerve conduction measurement lasts about 10 minutes.

After the patients surgery we will do genetic testing of MTHFR genotype.

All study samples have been collected.

Of note: there were no secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for elective surgery with expected duration > 2 hours
* Healthy patients undergoing moderate surgery where the use of N2O is unproblematic

Exclusion Criteria:

* Contraindication against N2O (pneumothorax, mechanical bowel obstruction, middle ear occlusion, laparoscopic surgery, raised intracranial pressure)
* Patients requiring supplemental oxygen
* Urgent or emergent surgery
* Patients with vitamin B12 or folate deficiency or megaloblastic anemia
* Patients with seizure disorder (epilepsy)
* Allergy or hypersensitivity against IV cobalamin or folate
* Patients with Leber's disease (hereditary optic nerve atrophy)
* Patients taking supplemental vitamin B12 or folate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nagele, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagele P, Zeugswetter B, Wiener C, Burger H, Hupfl M, Mittlbock M, Fodinger M. Influence of methylenetetrahydrofolate reductase gene polymorphisms on homocysteine concentrations after nitrous oxide anesthesia. Anesthesiology. 2008 Jul;109(1):36-43. doi: 10.1097/ALN.0b013e318178820b. PMID 18580170
- [Background] Nagele P, Zeugswetter B, Eberle C, Hupfl M, Mittlbock M, Fodinger M. A common gene variant in methionine synthase reductase is not associated with peak homocysteine concentrations after nitrous oxide anesthesia. Pharmacogenet Genomics. 2009 May;19(5):325-9. doi: 10.1097/FPC.0b013e328328d54c. PMID 19339913
- [Background] Myles PS, Chan MT, Kaye DM, McIlroy DR, Lau CW, Symons JA, Chen S. Effect of nitrous oxide anesthesia on plasma homocysteine and endothelial function. Anesthesiology. 2008 Oct;109(4):657-63. doi: 10.1097/ALN.0b013e31818629db. PMID 18813045

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 63 patients were consented however only 59 were analyzed.
Groups:
- B-vitamins Plus Nitrous Oxide: IV vitamin B12 (cyanocobalamin) 1 mg,
  IV folic acid, 5 mg,
  60% nitrous oxide
- Nitrous Oxide Plus Placebo: 60% nitrous oxide
  Placebo: normal saline (no vitamins)
- Nitrous Oxide-free Group Plus Placebo: No nitrous oxide during anesthesia (oxygen/nitrogen)
  Placebo: normal saline
Period: Overall Study
Arm/Group | B-vitamins Plus Nitrous Oxide | Nitrous Oxide Plus Placebo | Nitrous Oxide-free Group Plus Placebo
Started | 21 | 20 | 22
Completed | 20 | 19 | 20
Not Completed | 1 | 1 | 2
Not completed — Physician Decision | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | B-vitamins Plus Nitrous Oxide | Nitrous Oxide Plus Placebo | Nitrous Oxide-free Group Plus Placebo | Total
Number analyzed (Participants) | 20 | 19 | 20 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (13) | 40 (14) | 42 (15) | 41 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 12 | 33
  Male | 9 | 9 | 8 | 26
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 20 | 59

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Total Homocysteine Concentration (tHcy)
Description: Difference between baseline (pre-operative) and peak postoperative (i.e., maximum of postoperative value obtained within 30 minutes after anesthesia end time and morning of post-operative day 1) tHcy concentration .
  Of note: there were no secondary outcomes.
Time Frame: Immediately postoperatively and on postoperative day 1
Measure: Median (95% Confidence Interval); unit: mcmol/L
Groups:
- Treatment 1: B12-Folic acid, nitrous oxide
  B12-Folic Acid, nitrous oxide: IV vitamin B12 (cyanocobalamin) 1 mg, single administration over 30 min.
  IV folic acid, 5 mg, single administration over 30 min.
  Both diluted in 250 ml normal saline.
  Nitrous oxide (NO) and placebo: 60% nitrous oxide anesthesia plus saline
Arm/Group | Treatment 1 | Treatment 2 | Control Group
Number analyzed (Participants) | 20 | 19 | 20
mcmol/L | 1.9 [0.2 to 3.6] | 2.7 [0.6 to 4.8] | 0.5 [-0.8 to 1.9]
Statistical Analysis 1: Comparison: Treatment 1 vs Treatment 2 vs Control Group; For baseline comparisons among the three groups, one-way ANOVA was used for normally distributed variables and χ2 goodness-of-fit for categorical variables. To model the effects of B-vitamin treatment on nitrous-oxide-induced total homocysteine increase at the three different timepoints within individual patients and between the three groups, a linear mixed model with was used and we included a group × time interaction in the model; Test type: Superiority; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: AEs were assessed only in the immediate study period (surgery to postoperative day 1)
Arm/Group | B-vitamins Plus Nitrous Oxide | Nitrous Oxide Plus Placebo | Nitrous Oxide-free Group Plus Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 2/19 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B-vitamins Plus Nitrous Oxide (N=20) | Nitrous Oxide Plus Placebo (N=19) | Nitrous Oxide-free Group Plus Placebo (N=20)
PONV (Nervous system disorders) | 0 | 2 | 0 — Postopertaive nausea and vomiting
Postop. cardiac troponin elevation (Cardiac disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No